CLINICAL TRIAL: NCT06810843
Title: Sedation of Remazolam in Combination With Afentanil in Non-intubated Thoracoscopic Pulmonary Surgery: a Single-blind, Randomized, Controlled Trial
Brief Title: Sedation of Remazolam Combined With Afentanil in Non-intubated Thoracoscopic Pulmonary Surgery
Acronym: R-A NITS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Wu, chief physician, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YXLL-KY-2024(169)
Record Dates: First submitted 2025-01-18; First posted 2025-02-06 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Nodule Cm
Keywords: Non-intubated thoracoscopic surgery; Tubleless VATS; Remazolam; alfentanyl; NITS

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-R (Experimental): Afentanil (dose 10 μg/kg, Yichang Renfu Pharmaceutical Co., LTD.), 3 minutes before sedative administration. Then, in the remazolam group (group R), 0.3mg/kg remazolam (Yichang Renfu Pharmaceutical Co., LTD.) > 60 seconds. Sedation was maintained by continuous infusion of remazolam 0.2 to 1 mg/kg/h and afentanil 0 to 1μg/kg/min.
  Interventions: Drug: Remazolam combined with afentanil for non-intubated thoracoscopic surgery
- Group-P (Active Comparator): Propofol group (Group P) was given 1.5 to 2mg/kg propofol, continued infusion of propofol 2 to 6 mg/kg/h and afentanil 0 to 1μg/kg/min to maintain sedation. The anesthesiologist maintained sedation at the target level, maintaining the Modified Observer Alertness/Sedation Scale (MOAA/S) between 1-2.
  Interventions: Drug: Propofol combined with afentanil in non-intubated thoracoscopic surgery

INTERVENTIONS:
Drug: Remazolam combined with afentanil for non-intubated thoracoscopic surgery — Remazolam combined with afentanil for sedation in patients undergoing non-intubated thoracoscopic surgery,
  Other Names: Under the guidance of local anesthesia ultrasound, three paravertebral T4-5-6 points were blocked successively
  Arms: Group-R
Drug: Propofol combined with afentanil in non-intubated thoracoscopic surgery — Propofol combined with afentanil for sedation in patients undergoing non-intubated thoracoscopic surgery,
  Other Names: Under the guidance of local anesthesia ultrasound, three paravertebral T4-5-6 points were blocked successively
  Arms: Group-P

SUMMARY:
Non-intubated Thoracoscopic surgery (NITS) is a newly emerging minimally invasive surgical technique in recent years . Compared with traditional intubation general anesthesia, it has the advantages of less trauma, faster recovery and fewer complications . This surgical method allows patients to perform under local anesthesia or regional block and moderate sedation, providing a physiologic ventilation method , reducing the intervention on the respiratory system and conducive to rapid postoperative recovery.

The importance of sedative drugs in non-intubated thoracoscopic surgery Successful implementation of non-intubated thoracoscopic surgery requires sound regional block, airway management, and rational use of intravenous sedation and analgesics . In addition, sedative drugs need to have less respiratory and circulatory inhibition and fewer side effects. Propofol, as the most commonly used sedative drug, has a high incidence of adverse reactions such as injection pain and respiratory and circulatory inhibition. A large number of meta-analyses and systematic reviews have compared the sedative effects of remazolam and propofol, proving that Remazolam, as a new sedative, has advantages such as short half-life, rapid onset, rapid recovery, and light respiratory and circulatory inhibition.Compared with traditional benzodiazepines, Remazolam has a shorter half-life, which is conducive to rapid postoperative wakeup and reduces the risk of discomfort and cognitive dysfunction in patients. In addition, remazolam has little influence on the respiratory system and is relatively stable on the circulatory system ，which is an ideal sedation option for non-intubated thoracoscopic surgery that retains spontaneous respiration. Afentanil mainly acts on μ opioid receptors , and its analgesic intensity is about 15 times that of morphine, which has the advantages of rapid onset, short duration of action, rapid recovery, high safety, and few adverse reactions . Afentanil has a short half-life , mild respiratory depression, low incidence of cough, postoperative nausea and vomiting . Remazolam combined with afentanil is widely used in various surgeries or examinations that preserve spontaneous breathing, such as gastroenteroscopy, ERCP, hysteroscopy, short-term plastic surgery and fiberbronchoscopy, and has shown the advantage of light respiratory circulation inhibition . We speculate that remazolam combined with afentanil may have certain advantages in non-intubated thoracoscopic surgery that retains spontaneous breathing. At present, the application of remazolam combined with afentanil in non-intubated thoracoscopic surgery is still lacking. The purpose of this study was to observe the safety and effectiveness of remazolam combined with afentanil in non-intubated thoracoscopic surgery, and to provide a better choice of sedation drugs for non-intubated thoracoscopic surgery.

DETAILED DESCRIPTION:
Research object Patients aged 18 years or older undergoing non-intubated thoracoscopic lung surgery 3.2 Sample size calculation According to the study of Goyal R etal., propofo-based sedation resulted in a decrease in oxygen saturation in nearly 43% of patients. Therefore, assuming a 15% reduction in anoxic events in the remazolam group, PASS-2021 software, comparison of two independent sample rates, bilateral Z test, 80% confidence, and a significant difference level of 0.05, we estimated that the sample size in each group in this study was 156 patients, and considering the 20% shedding rate, 195 patients were required in each group. A sample size of 390 cases is required.

3.3 Scheduling Standards 3.3.1 Inclusion criteria:

1. American Society of Anesthesiologists ASA Level I to III;
2. 18 years old ≤ age ≤80 years old;
3. Non-intubated thoracoscopic lung surgery under deep sedation;
4. 18kg/m2≤BMI≤30 kg/m2;
5. Voluntarily participate in the study and sign the informed consent. 3.3.2 Exclusion criteria:

(1) Pulmonary function examination showed moderate to severe ventilation or exchange impairment (FEV1< 60% of the predicted value, carbon monoxide diffusion < 60% of the predicted value); (2) Abnormal liver and kidney function (Child-Pugh grade liver function is grade B and grade C; Endogenous creatinine clearance ≤50mL/min, serum creatinine >178µmol/L or renal function test urea nitrogen >9mmol/L) (3) SpO2 < 95% before operation; (4) History of recovery from abnormal surgical anesthesia; (5) History of thoracic surgery or history of tuberculosis or systemic infection within one month; (6) Severe cardiovascular and cerebrovascular diseases (patients with severe cardiovascular and cerebrovascular diseases: high risk of hypertension, untreated coronary heart disease, valvular heart disease, previous myocardial infarction, cerebral infarction, cerebral thrombus, cerebral hemorrhage); (7) Take monoamine oxidase inhibitors or antidepressants within 15 days; (8) Chronic pain from long-term use of analgesics or psychotropic drugs, alcoholism; (9) Known drug allergy; (10) expected difficult airway; (11) Pregnant women or women giving birth; (12) Participation in other drug trials within three months or inability to communicate well with researchers.

3.3.3 Shedding cases After signing informed consent and screening qualified for clinical trial, the patients did not complete the full clinical trial visit. Such as adverse events, patient loss of follow-up, patients who were converted to general anesthesia during the operation for reasons other than severe hypoxia, patients who could not complete the evaluation after surgery, patients voluntarily withdrew informed consent, and emergency blinding was initiated.

3.4 Randomization and blind method Block randomization was employed. The randomization scheme was generated by the researchers using the website (www.random.org). Random number in a light-tight sealed envelope. In this study, patients meeting the inclusion/exclusion criteria will be randomized into the trial group (remazolam, group R) and the control group (propofol, group P) in a 1:1 ratio. Since propofol is colored and remazolam is colorless, the anesthesiologist performing the anesthesia is non-blind. Follow-up personnel and statisticians, patients and chest doctors were blind.

3.5 Specific research content BIS, electrocardiogram, SpO2, blood pressure, heart rate, open venous access, nasal catheter oxygen inhalation (3L/min) were monitored. Under the guidance of local anesthesia ultrasound, three paravertebral T4-5-6 points were blocked successively, and 0.25% ropivacaine 15ml was administered. After disinfection, the anesthetic plane was tested to be effective before cutting the skin, then intravenous medication was started. If the patient is in pain before the incision, the surgeon gives additional local anesthesia and then starts intravenous medication. Two anesthesiologists are in charge of the patient throughout the procedure. Afentanil (dose 10μg/kg, Yichang Renfu Pharmaceutical Co., LTD.), 3 minutes before sedative administration. Then, in the remazolam group, 0.3mg/kg remazolam (Yichang Renfu Pharmaceutical Co., LTD.) was administered for > 60 seconds. Sedation was maintained by continuous infusion of remazolam 0.2 to 1mg/kg/h and afentanil 0 to 1μg/kg/min. The propofol group was given 1.5 to 2mg/kg propofol, continued infusion of propofol 2 to 6 mg/kg/h and afentanil 0 to 1μg/kg/min to maintain sedation. The anesthesiologist maintained sedation at the target level, maintaining the Modified Observer Alertness/Sedation Scale (MOAA/S) between 1-2. For example, if the MOAA/ S is higher than 2 and the patient is still overreacting and cannot tolerate surgery, use 0.1mg/kg remazolam push or 0.5mg/kg propofol, respectively, as additional sedation. In addition, both groups were given 5μg/kg of afentanil for additional analgesia. After surgery, patients were transferred to the recovery room, where their HR, SpO2, NIBP, and MOAA/S were monitored. A modified Aldrete score was used to assess recovery. Patients are only allowed to return to the room if their Aldrete score is at least 9 and there are no obvious side effects such as nausea or dizziness.

Hypotension was defined as MAP<65 mmHg or a 20% decrease from baseline, while hypertension was defined as MAP>105 mmHg or a 20% increase from baseline. According to the American Heart Association, when hypotension or hypertension occurs, we take two blood pressure readings immediately to provide a more accurate blood pressure. Patients with hypotension and accelerated heart rate received a 4ug norepinephrine push injection, then titrated to BP and heart rate. In contrast, patients with hypotension and HR < 60 bpm received a push dose of 10 mg ephedrine, which was then titrated to blood pressure and heart rate. In hypertensive patients, 5 mg urapidil was administered and titrated to BP. If the heart rate drops to <45 bpm, atropine 0.25mg is injected intravenously and titrated to the heart rate. If heart rate >110 bpm, Esmolol (10 mg) is administered intravenously and titrated to heart rate.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists ASA Level I to III;
* 18 years-80 years old;
* Non-intubated thoracoscopic lung surgery under deep sedation;
* 18 kg/m2≤BMI≤30 kg/m2;
* Voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

* Pulmonary function tests showed moderate to severe ventilation or exchange disorders (FEV1< 60% of the predicted value, carbon monoxide diffusion < 60% of the predicted value);
* Abnormal liver and kidney function (Child-Pugh grade liver function is grade B and grade C; Endogenous creatinine clearance ≤50mL/min, serum creatinine >178µmol/L or urea nitrogen >9mmol/L by renal function test);
* SpO2 < 95% before operation;
* History of recovery from abnormal surgical anesthesia;
* History of thoracic surgery or history of tuberculosis or systemic infection within one month;
* Severe cardiovascular and cerebrovascular diseases (patients with severe cardiovascular and cerebrovascular diseases:

High risk of hypertension, untreated coronary heart disease, valvular heart disease, previous myocardial infarction, cerebral infarction, cerebral thrombus, cerebral hemorrhage);

* Take monoamine oxidase inhibitors or antidepressants within 15 days;
* Chronic pain from long-term use of analgesics or psychotropic drugs, alcoholism;
* Known drug allergy;
* Expected difficult airway;
* Pregnant women or women giving birth;
* Participation in other drug trials within three months or inability to communicate well with researchers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of hypoxia | during the surgery
  The primary indicator was the incidence of hypoxia, defined as SpO2 < 90%,T>10s.Record whether and how often patients experienced pulse oxygen saturation below 90%.

SECONDARY OUTCOMES:
Frequency of intraoperative hypoxemia | during the surgery
  The frequency of intraoperative hypoxemia and the number of minor airway operations required and remedial measures such as jaw lift, increased oxygen flow, patient posture adjustment, mask ventilation, or endotracheal intubation during severe hypoxia. The minimum SpO2 and the number of assisted or mechanical ventilation due to hypoxia during the procedure were recorded. The occurrence of SpO2 < 90% was recorded.
the number of minor airway operations required and remedial measures | during the surgery
  The frequency of intraoperative hypoxemia and the number of minor airway operations required and remedial measures such as jaw lift, increased oxygen flow, patient posture adjustment, mask ventilation, or endotracheal intubation during severe hypoxia. The minimum SpO2 and the number of assisted or mechanical ventilation due to hypoxia during the procedure were recorded. The occurrence of SpO2 < 90% was recorded.
The minimum SpO2 were recorded | during the surgery
  The frequency of intraoperative hypoxemia and the number of minor airway operations required and remedial measures such as jaw lift, increased oxygen flow, patient posture adjustment, mask ventilation, or endotracheal intubation during severe hypoxia. The minimum SpO2 and the number of assisted or mechanical ventilation due to hypoxia during the procedure were recorded. The occurrence of SpO2 < 90% was recorded.
MAP at different time points | preinduction（T0） ,1minute （T1）、 3 minutes after induction（T2） ， At the beginning of the operation (T3)， 5 、10、15minutes after the operation began (T4、T5、T6) ，5minutes after withdrawal of anesthesia (T7)
  MAP at different time points were recorded
HR at different time points | preinduction（T0） ,1minute （T1）、 3 minutes after induction（T2） ， At the beginning of the operation (T3)， 5 、10、15minutes after the operation began (T4、T5、T6) ，5minutes after withdrawal of anesthesia (T7)
  HR at different time points were recorded
SpO2 at different time points | preinduction（T0） ,1minute （T1）、 3 minutes after induction（T2） ， At the beginning of the operation (T3)， 5 、10、15minutes after the operation began (T4、T5、T6) ，5minutes after withdrawal of anesthesia (T7)
  SpO2 at different time points were recorded
BIS at different time points | preinduction（T0） ,1minute （T1）、 3 minutes after induction（T2） ， At the beginning of the operation (T3)， 5 、10、15minutes after the operation began (T4、T5、T6) ，5minutes after withdrawal of anesthesia (T7)
  BIS at different time points were recorded
Quality of Recovery Questionnaire (QOR-15) | The first day after surgery
  patients were interviewed using the 15-item Quality of Recovery Questionnaire (QOR-15).QoR-15 questionnaire, QoR-15 is a patient-reported outcome measurement validated to measure QoR after surgery and general anaesthesia. It ranges from 0 to 150, with a higher score indicating better recovery. Scoring standard: QoR is classified as excellent (QoR-15 > 135), good (122 ≤ QoR-15 ≤ 135), moderate (90 ≤ QoR-15 ≤ 121) or poor (QoR-15 <90).

CONTACTS AND LOCATIONS:
Overall Officials: jian Bo Wu, PH.D, Study Chair — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University（Qianfoshan Hospital, Shandong Province）, Jinan, China